CLINICAL TRIAL: NCT07302529
Title: The Effect of a Mixed Intervention Structured According to the Integrated Disaster Management System on Disaster Risk Perception, Disaster Attitude and Brief Resilience Among University Students
Brief Title: The Effect of a Mixed Intervention Structured According to the Integrated Disaster Management System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Necmettin Erbakan University (Other)
Responsible Party: Principal Investigator, Kübra Sultan Dengiz, Lecturer, RN, PhD., Necmettin Erbakan University
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2025/1159
Record Dates: First submitted 2025-09-30; First posted 2025-12-24 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2025-12

CONDITIONS: Integrated Disaster Management System; University Students; Disaster Risk Perception; Disaster Attitude; Psychological Resilience; Perception
Keywords: Integrated Disaster Management System; Disaster Risk Perception; Disaster Attitude; Psychological Resilience; University Students; Nursing

STUDY DESIGN:
Intervention Model Description: A 15-week mixed intervention will be implemented in the experimental group. The intervention will include lectures on disaster culture, conferences by Red Crescent staff and AKUT volunteers, case studies structured according to the integrated disaster management system, a disaster simulation application, and student material development.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Masking will be ensured in the study in terms of data/output measurement, statistical analysis and reporting. A psychological resilience scale was added as a measurement tool to mask the effect of the instrument.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention group (Experimental): Disaster culture course presentations, conferences by Red Crescent personnel and AKUT volunteers, and the integrated disaster management system were structured according to the; Case studies, disaster simulation application, and student material development will be included.
  Interventions: Behavioral: Mixed Intervention
- Control group (No Intervention): no intervention will be implemented.

INTERVENTIONS:
Behavioral: Mixed Intervention — This study is distinguished by the fact that the intervention was conducted on university students, the intervention was structured according to the integrated disaster management system, case studies and simulation were included in the training content, conferences by field professionals in disaster management were included in the initiative, and the study team consisted of doctoral-level researchers.
  Arms: intervention group

SUMMARY:
Integrated disaster management is defined as a management process that considers all hazards to create a resilient and resilient society capable of coping with disasters, and utilizes all the resources and resources of society to implement the necessary actions and measures in the prevention, mitigation, preparedness, response, and recovery phases of disaster management. Educational interventions for disaster management are the most important initiatives in both risk reduction and crisis management. In this context, the aim of this study is to evaluate the impact of a hybrid intervention structured according to the integrated disaster management system on disaster risk perception, disaster attitudes, and psychological resilience in university students. The students participating in this study will be administered a mixed intervention structured according to the integrated disaster management system (15-week disaster culture course presentation, case studies, simulation, expert conferences, and material development). Because randomization is not possible, the study adopts a quasi-experimental design. However, measures will be taken to reduce the risk of bias by creating a control group, increasing the number of measurements, using a different scale for test measurements, and ensuring that the individuals implementing the interventions, performing data analysis, and performing the measurements are different. The disaster risk perception scale, disaster attitude scale, and brief psychological resilience scale will be used to collect data. Data analysis will be evaluated at a 95% confidence interval and a significance level of p<0.05.

ELIGIBILITY:
Inclusion Criteria:

* Registered as a student at the university where the research will be conducted
* Active participation in the disaster culture course

Exclusion Criteria:

* There are no exclusion criteria.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2025-10-31 (Actual); Primary Completion 2025-12-25 (Actual); Study Completion 2026-02-10 (Actual)

PRIMARY OUTCOMES:
disaster risk perception | From enrollment to the end of treatment at 15 weeks
  Changes disaster risk perception scores after a structured mixed intervention based on an integrated disaster management system implemented on university students
disaster attitude | From enrollment to the end of treatment at 15 weeks
  Changes disaster attitude scores after a structured mixed intervention based on an integrated disaster management system implemented on university students

SECONDARY OUTCOMES:
psychological resilience | From enrollment to the end of treatment at 15 weeks
  Changes psychological resilience scores after a structured mixed intervention based on an integrated disaster management system implemented on university students

CONTACTS AND LOCATIONS:
Locations (1):
- Necmettin Erbakan University, Faculthy of Nursing, Konya, Konya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No